CLINICAL TRIAL: NCT00101660
Title: A Phase II Study to Determine the Activity of BMS-354825 in Subjects With Chronic Phase Philadelphia Chromosome-Positive Chronic Myeloid Leukemia Who Have Disease That is Resistant to High Dose Imatinib Mesylate (Gleevec) or Who Are Intolerant of Imatinib
Brief Title: Study of BMS-354825 (Dasatinib) in Patients With Chronic Myeloid Leukemia Who Are Either Resistant or Intolerant to Imatinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-013; NCT00112801 (obsolete NCT alias)
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Results first posted 2010-02-24 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Myeloid Leukemia; Philadelphia-Positive Myeloid Leukemia
Keywords: Chronic phase Philadelphia chromosome chronic myeloid leukemia (Ph+CML)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib, 70 mg twice daily (BID) (Experimental): Dasatanib, 70 mg twice daily (BID), with dose escalation to 90 mg BID was allowed for participants who showed evidence of progression or lack of response. Up to 2 dose reductions were allowed for intolerance.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets; oral; 70 mg BID, depending on response

SUMMARY:
The purpose of this study is assess the effects of the investigational drug dasatinib on participants who are in chronic phase Philadelphia chromosome chronic myeloid leukemia and who are either resistant to or intolerant of imatinib. Other purposes of the study are to identify any side effects the drug may produce and to study the level of dasatanib in the blood and assess the efficacy of dasatanib in the treatment of leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and older.
* Chronic myeloid leukemia (CML)
* Previous treatment with imatinib at a dose of >600 mg/day AND the development of progressive disease while receiving imatinib at that dose, OR
* CML with resistance to imatinib at a dose less than or equal to 600 mg/day with genetic mutation in the BCR-ABL gene that is associated with a high level of resistance to imatinib, OR
* Intolerance to imatinib at any dose
* Adequate organ function
* Women who are able to bear children must have a negative serum or urine pregnancy test. Adequate methods of contraception must be used throughout the study to avoid pregnancy for the entire interval of at least 1 month before and 3 months after completion of the study medication.

Exclusion Criteria:

* Woman who are pregnant or breastfeeding
* Men whose sexual partners are women who are of childbearing potential, and who are unwilling or unable to use an acceptable method to avoid pregnancy of his partner for the entire study period as outlined above
* Previous diagnosis of accelerated phase or blast crisis CML.
* Participants who are eligible and willing to undergo transplantation during the screening period
* Uncontrolled or significant cardiovascular disease
* Use of imatinib within 7 days.
* Use of interferon or cytarabine within 14 days
* Use of a targeted small-molecule anticancer agent within 14 days
* Use of certain medication that carry a known side effect risk of Torsade de Pointes - Certain medications that irreversibly inhibit platelet function or anticoagulants
* Prior therapy with dasatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2005-02; Primary Completion 2006-09 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (85):
- United States (32):
  - Local Institution, Anaheim, California
  - Local Institution, Loma Linda, California
  - Local Institution, Los Angeles, California
  - Local Institution, Stanford, California
  - Local Institution, Vallejo, California
  - Local Institution, Hartford, Connecticut
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Jacksonville, Florida
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Kansas City, Kansas
  - Local Institution, Baltimore, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Detroit, Michigan
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Omaha, Nebraska
  - Local Institution, Hackensack, New Jersey
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, New York, New York
  - Local Institution, Portland, Oregon
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Greenville, South Carolina
  - Local Institution, Nashville, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Tyler, Texas
  - Local Institution, Spokane, Washington
- Australia (5):
  - Local Institution, St Leonards, New South Wales
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, East Mebourne, Victoria
  - Local Institution, Parkville, Victoria
- Local Institution, Wein, Austria
- Belgium (4):
  - Local Institution, B-Leuven
  - Local Institution, Brussels
  - Local Institution, Edegem
  - Local Institution, Yvoir
- Canada (3):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- Local Institution, Aarhus, Denmark
- Local Institution, Helsinki, Finland
- France (7):
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (4):
  - Local Institution, Hamburg
  - Local Institution, Leipzig
  - Local Institution, Mainz
  - Local Institution, Mannheim
- Ireland (2):
  - Local Institution, Co Galway, Galway
  - Local Institution, Dublin
- Local Institution, Ramat Gan, Israel
- Italy (6):
  - Local Institution, Bari
  - Local Institution, Bologna
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Orbassano
  - Local Institution, Roma
- Netherlands (2):
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
- Local Institution, Trondheim, Norway
- Local Institution, Lima, Lima Province, Peru
- Local Institution, Singapore, Singapore
- South Africa (2):
  - Local Institution, Parktown, Gauteng
  - Local Institution, Soweto, Gauteng
- Local Institution, Kyunggi-Do, South Korea
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Sweden (5):
  - Local Institution, Gothenburg
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Umeå
  - Local Institution, Uppsala
- Local Instituion, Basel, Switzerland
- United Kingdom (2):
  - Local Institution, Glasgow, Central
  - Local Institution, London, Greater London

REFERENCES:
- [Background] Hochhaus A, Kantarjian HM, Baccarani M, Lipton JH, Apperley JF, Druker BJ, Facon T, Goldberg SL, Cervantes F, Niederwieser D, Silver RT, Stone RM, Hughes TP, Muller MC, Ezzeddine R, Countouriotis AM, Shah NP. Dasatinib induces notable hematologic and cytogenetic responses in chronic-phase chronic myeloid leukemia after failure of imatinib therapy. Blood. 2007 Mar 15;109(6):2303-9. doi: 10.1182/blood-2006-09-047266. Epub 2006 Nov 30. PMID 17138817
- [Background] Muller MC, Cortes JE, Kim DW, Druker BJ, Erben P, Pasquini R, Branford S, Hughes TP, Radich JP, Ploughman L, Mukhopadhyay J, Hochhaus A. Dasatinib treatment of chronic-phase chronic myeloid leukemia: analysis of responses according to preexisting BCR-ABL mutations. Blood. 2009 Dec 3;114(24):4944-53. doi: 10.1182/blood-2009-04-214221. Epub 2009 Sep 24. PMID 19779040

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib-intolerant: Imatinib intolerance was defined as: Grade 3 or greater nonhematologic toxicity that is imatinib-related or Grade 4 hematologic toxicity that is imatinib-related lasting more than 7 days.
- Imatinib-resistant: Imatinib resistance, acquired or primary. Acquired resistance: participants who achieve major cytogenetic response (MCyR) or complete hematologic response (CHR) on imatinib at any dose prior to progression, defined by 1 of the following: loss of MCyR, loss of CHR, or increasing white blood cell (WBC) count. Primary resistance: participants who never achieve MCyR or CHR at any dose, and meet 1 of the following: continuously increasing WBC count on at least 2 consecutive evaluations at least 2 weeks apart, with the final assessment showing a doubling of WBC from nadir to ≥20,000/mm^3; an absolute increase in WBC by more than 50,000/mm^3 above lowest count after starting imatinib; no CHR after 3 months; no cytogenetic response (CyR) after 6 months; or no MCyR after 12 months. Resistance was also defined as chronic myeloid leukemia (CML) with resistance to imatinib ≤600mg/d with genetic mutation in BCR-ABL gene (L248V, G250E, Q252H/R, Y253H/F, E255K/V, T315I/D, F317L, H369P/R).
Period: Overall Study
Arm/Group | Imatinib-intolerant | Imatinib-resistant
Started | 99 | 288
Completed | 99 | 288
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib-intolerant | Imatinib-resistant | Total
Number analyzed (Participants) | 99 | 288 | 387
Age Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (12.5) | 55.7 (13.5) | 55.4 (13.3)
Age, Customized [Number; unit: Participants]
  Between 21 and 45 years | 25 | 78 | 103
  Between 46 and 65 years | 55 | 131 | 186
  Between 66 and 75 years | 17 | 65 | 82
  > 75 years | 2 | 14 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 139 | 196
  Male | 42 | 149 | 191
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 93 | 252 | 345
  Black/African American | 2 | 13 | 15
  Asian | 3 | 10 | 13
  Other | 1 | 12 | 13
  Not reported | 0 | 1 | 1
Performance Status - Eastern Cooperative Oncology Group Scale (ECOG) Score [Number; unit: Participants] — ECOG scale is a 6-item scale used to assess disease progression, daily functioning, and appropriate treatment and prognosis. Scale 1-5, with 0=fully active, able to carry on all predisease performance without restriction, 1=physically strenous activity restricted, 2=capable of self-care, unable to work, 3=capable of only limited self-care, bed/chair confined for >50% of time, 4=completely disbled, bed/chair confined, and 5=death
  Participants
    0 | 71 | 205 | 276
    1 | 28 | 77 | 105
    2 | 0 | 3 | 3
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0
    Not reported | 0 | 3 | 3
Functional Assessment of Cancer Therapy-General (FACT-G) [Mean (Standard Deviation); unit: Units on a scale] — FACT-G=27 questions in 4 domains: physical, social/family, emotional, functional well-being (PWB, SWB, EWB, FWB). Total score=0 to 108; higher score=better health-related quality of life. 13 participants in imatinib-intolerant group had baseline measurements; 161 participants in imatinib-resistant group had baseline measurements for all 4 domains/79 had baseline measurements for total scores. Imatinib-intolerant participants assessed at baseline: n=78 for Total, EWB, FWB; n=80 for PWB, SWB. Imatinib-resistant participants assessed at baseline: n=234, Total; n=238, PWB, FWB; n=237, SWB, EWB.
  Units on a scale
    Total FACT-G | 81.1 (14.4) | 82.4 (13.1) | 82.1 (13.4)
    PWB | 22.0 (5.1) | 21.6 (5.2) | 21.7 (5.2)
    SWB | 23.0 (4.4) | 23.0 (4.5) | 23.0 (4.4)
    EWB | 17.3 (4.0) | 18.4 (3.7) | 18.1 (3.8)
    FWB | 18.7 (5.5) | 19.6 (5.6) | 19.4 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Imatinib-resistant Participants With Major Cytogenetic Response (MCyR)
Description: Cytogenetic response was based on the prevalence of Ph+ metaphases among cells with metaphases in a bone marrow sample. MCyR is the combination of Complete Cytogenetic Response (CCyR)-0% Ph+ metaphases plus Partial Cytogenetic Response (PCyR)-1% to 35% Ph+ metaphases.
Time Frame: 2 years
Population: All imatinib-resistant participants who received treatment.
Measure: Number; unit: Participants
Groups:
- Dasatinib, 70 mg, Twice Daily (BID): Dasatinib, 70 mg BID, with dose escalation to 90 mg BID was allowed for participants who showed evidence of progression or lack of response. Up to 2 dose reductions were allowed for intolerance.
Arm/Group | Dasatinib, 70 mg, Twice Daily (BID)
Number analyzed (Participants) | 288
Participants | 159

2. Secondary Outcome: Number of Imatinib-intolerant Participants With MCyR
Description: Determination of cytogenetic response was based on the prevalence of Ph+ metaphases among cells with metaphases in a bone marrow sample. MCyR is the combination of CCyR-0% Ph+ metaphases and PCyR - 1% to 35% Ph+ metaphases.
Time Frame: Baseline to 2 years
Population: All imatinib-intolerant participants who received treatment.
Measure: Number; unit: Participants
Groups:
- Dastinib, 70 mg, BID: Dasatinib, 70 mg BID, with dose escalation to 90 mg BID was allowed for participants who showed evidence of progression or lack of response. Up to 2 dose reductions were allowed for intolerance.
Arm/Group | Dastinib, 70 mg, BID
Number analyzed (Participants) | 99
Participants | 81

3. Secondary Outcome: Percentage of Participants Who Achieved MCyR and Did Not Progress at 12 and 24 Months
Description: Based on the Kaplan-Meier estimate of the duration of response. Determination of cytogenetic response was based on the prevalence of Ph+ metaphases among cells with metaphases in a bone marrow sample. MCyR is the combination of Complete Cytogenetic Response (CCyR)-0% Ph+ metaphases and Partial Cytogenetic Response (PCyR) - 1% to 35% Ph+ metaphases.
Time Frame: 12 and 24 Months
Population: Population is limited to responders (those who acheived MCyR) who were also assessed for duration of MCyR.
Measure: Number; unit: Percentage of participants
Groups:
- Dasatanib, 70 mg BID: Dasatinib, 70 mg BID, with dose escalation to 90 mg BID was allowed for participants who showed evidence of progression or lack of response. Up to 2 dose reductions were allowed for intolerance.
Arm/Group | Dasatanib, 70 mg BID
Number analyzed (Participants) | 240
Percentage of participants
  Imatinib-intolerant group: 12 months (n=81) | 98.5
  Imatinib-intolerant group: 24 months (n=81) | 96.7
  Imatinib-resistant group: 12 months (n=159) | 93.7
  Imatinib-resistant group: 24 months (n=159) | 83.6

4. Secondary Outcome: Median Time From First Dosing Date to Date of MCyR
Description: MCyR is the combination of CCyR-0% Ph+ metaphases and PCyR - 1% to 35% Ph+ metaphases.
Time Frame: Baseline (within 4 weeks of Day 1) and every 12 weeks
Population: Population is limited to responders (those who acheived MCyR) only
Measure: Median (Full Range); unit: Months
Groups:
- Dasatinib, 70 mg BID: Dasatinib, 70 mg BID, with dose escalation to 90 mg BID was allowed for participants who showed evidence of progression or lack of response. Up to 2 dose reductions were allowed for intolerance.
Arm/Group | Dasatinib, 70 mg BID
Number analyzed (Participants) | 240
Months
  Imatinib-intolerant | 2.79 [0.79 to 16.39]
  Imatinib-resistant | 2.92 [0.95 to 22.37]

5. Secondary Outcome: Number of Participants With Complete Hematologic Response (CHR)
Description: CHR=all of the following criteria: white blood cell count ≤ institutional upper limit of normal; platelets <450,000/mm^3; no blasts or promyelocytes in peripheral blood; <5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils ≤20%; no extramedullary involvement. Response, as defined, must be maintained for at least 4 weeks after first documented. A CHR could begin only 14 days after dosing start date.
Time Frame: Baseline (within 72 hours of start of therapy), weekly until Week 12, every 3 months until off-study
Population: All participants who received treatment.
Measure: Number; unit: Participants
Groups:
- Dasatinib, 70 mg BID: Dasatinib, 70 mg twice BID, with dose escalation to 90 mg BID was allowed for participants who showed evidence of progression or lack of response. Up to 2 dose reductions were allowed for intolerance.
Arm/Group | Dasatinib, 70 mg BID
Number analyzed (Participants) | 387
Participants
  Imatinib-intolerant (n=99) | 93
  Imatinib-resistant (n=288) | 259

6. Secondary Outcome: Percentage of Participants Who Acheived CHR and Did Not Progress at 12 Months and 24 Months
Description: Based on the Kaplan-Meier estimate of the duration of response. CHR=all of the following criteria: white blood cell count ≤ institutional upper limit of normal; platelets < 450,000/mm^3; no blasts or promyelocytes in peripheral blood; <5% myelocytes plus metamyelocytes in peripheral blood; peripheral blood basophils ≤20%; no extramedullary involvement. Response, as defined, must be maintained for at least 4 weeks after first documented. A CHR could begin only 14 days after dosing start date.
Time Frame: 12 and 24 months
Population: Population limited to responders (those achieving CHR) only
Measure: Number; unit: Percentage of participants
Groups:
- Dasatinib,70 mg BID: Dasatanib, 70 mg BID, with dose escalation to 90 mg BID was allowed for participants who showed evidence of progression or lack of response. Up to 2 dose reductions were allowed for intolerance.
Arm/Group | Dasatinib,70 mg BID
Number analyzed (Participants) | 352
Percentage of participants
  Imatinib-intolerant: 12 months (n=93) | 97.7
  Imatinib-intolerant: 24 months (n=93) | 93.5
  Imatinib-resistant: 12 months (n=259) | 90.4
  Imatinib-resistant: 24 months (n=259) | 78.8

7. Secondary Outcome: Median Time From First Dosing Until CHR
Description: as for outcome 5
Time Frame: Baseline (within 72 hours of start of therapy), weekly until Week 12, every 3 months until off-study
Population: Population limited to responders (those achieving CHR) only
Measure: Median (Full Range); unit: Months
Arm/Group | Dasatinib, 70 mg BID
Number analyzed (Participants) | 352
Months
  Imatinib-intolerant (n=93) | 0.49 [0.46 to 3.78]
  Imatinib-resistant (n=259) | 0.53 [0.46 to 12.39]

8. Secondary Outcome: Number of Participants With Major Molecular Response (MMR)
Description: MMR is defined as ≤3 log reduction in BCR-ABL levels from the standardized baseline value of BCR-ABL:Control Gene ratio. The international ratio is obtained by multiplying BCR-ABL:Control gene ratio by the lab-specific conversion factor.
Time Frame: Baseline to 2 years
Population: All participants who received treatment.
Measure: Number; unit: Participants
Arm/Group | Dasatinib, 70 mg BID
Number analyzed (Participants) | 387
Participants
  Imatinib-intolerant (n=99) | 73
  Imatinib-resistant (n=288) | 102

9. Secondary Outcome: Minimal Clinically Significant Change From Baseline in Functional Assessment of Cancer Therapy-General (FACT-G) Questionnaire Scores
Description: Health-related quality of life as measured by FACT-G, which comprises 27 questions in 4 domains: PWB, SWB, EWB, FWB. Total FACT-G score=summation of the 4 subscale scores and ranges from 0 to 108. Higher scores=better health-related quality of life. Total Score change of 7 or more=minimal clinical important change; PWB, EWB, & FWB score change of 3 or more, and SWB score change of 2 or more=minimal clinical important change. Baseline FACT-G measurements can be found in Baseline Characteristics.
Time Frame: Baseline, Day 29, every 4 weeks for the first 24 weeks, then every 12 weeks for the remainder of treatment, after end of treatment. Treatment continued until disease progression or development of toxicity or until other protocol-defined criteria.
Population: Number of participants with assessments at baseline and timepoint
Measure: Number; unit: Participants
Arm/Group | Dasatinib,70 mg BID
Number analyzed (Participants) | 321
Participants
  Imatinib-intolerant: Total FACT-G (n=80) | 34
  Imatinib-intolerant: PWB (n=80) | 36
  Imatinib-intolerant: SWB (n=80) | 33
  Imatinib-intolerant: EWB (n=80) | 40
  Imatinib-intolerant: FWB (n=80) | 32
  Imatinib-resistant: Total FACT-G (n=241) | 107
  Imatinib-resistant: PWB (n=241) | 103
  Imatinib-resistant: SWB (n=241) | 94
  Imatinib-resistant: EWB (n=241) | 107
  Imatinib-resistant: FWB (n=241) | 89

10. Secondary Outcome: Number of Imitanib-intolerant Participants With Drug-related Adverse Events (AEs), Death Within 30 Days of Last Dose, Death, and AEs Leading to Discontinuation, Serious Adverse Events (SAEs), Grade 3-4 Thrombocytopenia, Grade 4-4 Neutropenia, and Any AE
Description: AE=any new untoward medical occurrence or worsening of a preexisting medical condition regardless of causal relationship with treatment. SAE=any untoward medical occurrence at any dose that: results in death; is life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability; is cancer; is congenital anomaly/birth defect; results in drug dependency/abuse; is an important medical event. Graded by National Cancer Institute Common Terminology Criteria for Adverse Events v3.0. (1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death)
Time Frame: Continuously, from baseline through 2 years
Population: All imitanib-intolerant participants who received treatment.
Measure: Number; unit: Participants
Arm/Group | Dasatinib,70 mg BID
Number analyzed (Participants) | 99
Participants
  Drug-related AEs | 97
  Death within 30 days of last dose | 0
  Deaths | 0
  On-study AEs leading to discontinuation | 16
  SAEs | 48
  Grade 3-4 thrombocytopenia | 32
  Grade 3-4 neutropenia | 39
  Any AE | 98

11. Secondary Outcome: Number of Imitanib-resistant Participants With Drug-related AEs, Death Within 30 Days of Last Dose, Death, AEs Leading to Discontinuation, SAEs, Grade 3-4 Thrombocytopenia, Grade 3-4 Neutropenia, and Any AE
Description: as for outcome 10
Time Frame: Continuously, from baseline through 2 years
Population: All imitanib-resistant participants who received treatment.
Measure: Number; unit: Participants
Groups:
- Dasatinib,70 mg BID: Dasatinib, 70 mg BID, with dose escalation to 90 mg BID was allowed for participants who showed evidence of progression or lack of response. Up to 2 dose reductions were allowed for intolerance.
  a
Arm/Group | Dasatinib,70 mg BID
Number analyzed (Participants) | 288
Participants
  Drug-related AEs | 281
  Death within 30 days of last dose | 8
  Deaths | 19
  On-study AEs leading to Discontinuation | 53
  SAEs | 146
  Grade 3-4 thrombocytopenia | 156
  Grade 3-4 neutropenia | 154
  Any AE | 288

12. Secondary Outcome: Blood Sample Collection for Pharmacokinetic (PK) Analysis of Dasatinib
Description: Blood samples were collected for PK to be included in separate population PK analyses.
Time Frame: Day 8 of study; pretreatment through sample between 30 minutes and 3 hours following treatment, a sample between 5 hours and 8 hours following treatment and a sample at 12 hours, prior to the next dose.
Population: No study-specific PK analyses were planned for this report.
Measure: Number; unit: Participants
Groups:
- Dasatinib: Dasatanib, 70 mg BID, with dose escalation to 90 mg BID was allowed for participants who showed evidence of progression or lack of response. Up to 2 dose reductions were allowed for intolerance.
Arm/Group | Dasatinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Intolerant | Resistant
Serious Adverse Events (participants affected / at risk) | 48/99 | 146/288
Other Adverse Events (participants affected / at risk) | 96/99 | 287/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intolerant (N=99) | Resistant (N=288)
LIPASE (Investigations) | 1 | 0
PROLONGED (Investigations) | 0 | 0
PLEUROSCOPY (Investigations) | 0 | 1
PLATELET COUNT (Investigations) | 0 | 2
WEIGHT DECREASED (Investigations) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 2
BLOOD CULTURE POSITIVE (Investigations) | 0 | 1
BLOOD CREATINE INCREASED (Investigations) | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 1 | 2
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 1
BIOPSY BONE MARROW ABNORMAL (Investigations) | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 1
ELECTROCARDIOGRAM QT CORRECTED INTERVAL (Investigations) | 0 | 0
CYANOSIS (Cardiac disorders) | 0 | 1
NODAL RHYTHM (Cardiac disorders) | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1
PERICARDITIS (Cardiac disorders) | 1 | 1
CARDIOMYOPATHY (Cardiac disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 2 | 1
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 7
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 3
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 5 | 9
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 2
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 2 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
EMBOLISM (Vascular disorders) | 1 | 0
HAEMATOMA (Vascular disorders) | 0 | 2
HYPERTENSION (Vascular disorders) | 1 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1
GOITRE (Endocrine disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1
HYPERSENSITIVITY (Immune system disorders) | 1 | 2
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 1
DIZZINESS (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 2
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 1
ILEUS (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 2
COLITIS (Gastrointestinal disorders) | 1 | 1
MELAENA (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 3
DIARRHOEA (Gastrointestinal disorders) | 2 | 10
ENTERITIS (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 1
GINGIVITIS (Gastrointestinal disorders) | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 1
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 0
PERIODONTITIS (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 4
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 4
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 1
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 0 | 2
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
EAR HAEMORRHAGE (Ear and labyrinth disorders) | 0 | 1
INFECTION (Infections and infestations) | 0 | 3
INFLUENZA (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 5 | 11
BRONCHITIS (Infections and infestations) | 1 | 4
CELLULITIS (Infections and infestations) | 2 | 4
APPENDICITIS (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 2
PNEUMONIA FUNGAL (Infections and infestations) | 0 | 1
FEBRILE INFECTION (Infections and infestations) | 1 | 0
VIRAL PHARYNGITIS (Infections and infestations) | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1
PERIRECTAL ABSCESS (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1
HERPES VIRUS INFECTION (Infections and infestations) | 0 | 1
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
PHARYNGOLARYNGEAL ABSCESS (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 0 | 2
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
POLLAKIURIA (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 4
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 2
GLOMERULONEPHROPATHY (Renal and urinary disorders) | 0 | 1
HYSTERECTOMY (Surgical and medical procedures) | 0 | 1
BONE MARROW TRANSPLANT (Surgical and medical procedures) | 0 | 2
CORONARY ARTERIAL STENT INSERTION (Surgical and medical procedures) | 0 | 1
ANOREXIA (Metabolism and nutrition disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 3
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 2 | 6
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 8
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 7
ACNE (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 0 | 1
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 | 1
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 15
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 16 | 32
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 5
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NASAL SEPTUM DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 3 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PAIN (General disorders) | 0 | 1
DEATH (General disorders) | 0 | 1
FATIGUE (General disorders) | 0 | 3
MALAISE (General disorders) | 1 | 1
PYREXIA (General disorders) | 3 | 26
ASTHENIA (General disorders) | 0 | 1
CHEST PAIN (General disorders) | 1 | 2
ADVERSE EVENT (General disorders) | 1 | 0
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LEIOMYOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BLAST CRISIS IN MYELOGENOUS LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intolerant (N=99) | Resistant (N=288)
EYELID OEDEMA (Eye disorders) | 5 | 6
VISION BLURRED (Eye disorders) | 8 | 12
WEIGHT DECREASED (Investigations) | 12 | 39
WEIGHT INCREASED (Investigations) | 10 | 30
PALPITATIONS (Cardiac disorders) | 6 | 16
PERICARDIAL EFFUSION (Cardiac disorders) | 5 | 13
FLUSHING (Vascular disorders) | 9 | 14
HOT FLUSH (Vascular disorders) | 5 | 14
HYPERTENSION (Vascular disorders) | 9 | 19
ANXIETY (Psychiatric disorders) | 6 | 17
INSOMNIA (Psychiatric disorders) | 14 | 33
DEPRESSION (Psychiatric disorders) | 10 | 20
HEADACHE (Nervous system disorders) | 49 | 128
DIZZINESS (Nervous system disorders) | 17 | 56
DYSGEUSIA (Nervous system disorders) | 5 | 10
PARAESTHESIA (Nervous system disorders) | 7 | 33
NAUSEA (Gastrointestinal disorders) | 40 | 108
COLITIS (Gastrointestinal disorders) | 5 | 6
VOMITING (Gastrointestinal disorders) | 17 | 64
DIARRHOEA (Gastrointestinal disorders) | 44 | 153
DYSPEPSIA (Gastrointestinal disorders) | 13 | 19
TOOTHACHE (Gastrointestinal disorders) | 3 | 15
FLATULENCE (Gastrointestinal disorders) | 9 | 18
STOMATITIS (Gastrointestinal disorders) | 3 | 15
CONSTIPATION (Gastrointestinal disorders) | 8 | 54
HAEMORRHOIDS (Gastrointestinal disorders) | 11 | 17
ABDOMINAL PAIN (Gastrointestinal disorders) | 17 | 47
MOUTH ULCERATION (Gastrointestinal disorders) | 2 | 15
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 9 | 27
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 14 | 36
SINUSITIS (Infections and infestations) | 8 | 17
BRONCHITIS (Infections and infestations) | 8 | 23
ORAL HERPES (Infections and infestations) | 4 | 24
NASOPHARYNGITIS (Infections and infestations) | 17 | 53
URINARY TRACT INFECTION (Infections and infestations) | 4 | 19
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 19 | 36
ANOREXIA (Metabolism and nutrition disorders) | 16 | 52
ANAEMIA (Blood and lymphatic system disorders) | 12 | 33
NEUTROPENIA (Blood and lymphatic system disorders) | 16 | 52
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 12 | 67
ACNE (Skin and subcutaneous tissue disorders) | 12 | 17
RASH (Skin and subcutaneous tissue disorders) | 43 | 103
ALOPECIA (Skin and subcutaneous tissue disorders) | 15 | 24
DRY SKIN (Skin and subcutaneous tissue disorders) | 9 | 18
ERYTHEMA (Skin and subcutaneous tissue disorders) | 11 | 19
PRURITUS (Skin and subcutaneous tissue disorders) | 18 | 36
URTICARIA (Skin and subcutaneous tissue disorders) | 5 | 10
SKIN LESION (Skin and subcutaneous tissue disorders) | 9 | 18
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 7 | 34
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 | 17
PERIORBITAL OEDEMA (Skin and subcutaneous tissue disorders) | 13 | 28
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 7 | 9
CONTUSION (Injury, poisoning and procedural complications) | 5 | 21
MYALGIA (Musculoskeletal and connective tissue disorders) | 19 | 49
BACK PAIN (Musculoskeletal and connective tissue disorders) | 19 | 53
BONE PAIN (Musculoskeletal and connective tissue disorders) | 10 | 48
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 24
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 | 86
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 10 | 27
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 18 | 58
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 12 | 27
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 5 | 17
COUGH (Respiratory, thoracic and mediastinal disorders) | 36 | 110
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 46 | 128
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 5 | 9
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 5 | 7
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 27
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 9
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 37 | 90
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 5 | 21
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14 | 42
PAIN (General disorders) | 6 | 21
CHILLS (General disorders) | 10 | 31
OEDEMA (General disorders) | 2 | 15
FATIGUE (General disorders) | 48 | 136
PYREXIA (General disorders) | 33 | 104
ASTHENIA (General disorders) | 19 | 58
CHEST PAIN (General disorders) | 17 | 35
CHEST DISCOMFORT (General disorders) | 10 | 19
OEDEMA PERIPHERAL (General disorders) | 24 | 75
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.